CLINICAL TRIAL: NCT05188066
Title: Study of Pregnancy Pathologies Associated With Placental Abnormalities
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC20.115
Record Dates: First submitted 2021-12-18; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Pre-eclampsia; Pre-Term; Fetal Growth Retardation
Keywords: pre-eclampsia; fetal growth retardation; placenta histology; vascularization; trophoblast proliferation
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Fetal Growth Retardation; Neovascularization, Pathologic | interventions — Shadowing Technique, Histology; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placenta and fetal membrane from normal and pathological pregnancies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal, pathological IVG: We will use placenta and fetal memebranes collected from first trimester termination of pregnancy. This will constitute group IVG.
  Interventions: Diagnostic Test: Histology
- Normal and pathological term: We will also use the same specimens collected from third trimester pregnancies . We will call this group normal and pathological..... à finaliser
  Interventions: Diagnostic Test: Histology

INTERVENTIONS:
Diagnostic Test: Histology — Collect the placenta and fetal membranes and perfor either tissue culture or fixation for further analyses
  Other Names: immunohistochemistry

SUMMARY:
Pregnancy pathologies can occur from implantation until childbirth. The investigators are interested in the development mechanisms of these pathologies and aim to develop therapies to treat them.

The investigators need to collect samples, especially placental samples, following abortions and term and premature deliveries. Abortions will allow investigators to have non-pathological placental material up to 13 weeks. This material will serve as a reference for the understanding of the histological changes that occur in normal placentas collected at term of pregnancy. The latter will, in turn, be compared with the placentas collected during premature deliveries. Also, the abortion product will be cultivated in an environment mimicking the pathology of pre-eclampsia. This study will allow investigators to advance their understanding of the pathophysiological mechanisms of the placenta. The investigators are internationally recognized for their research on these pathologies.

DETAILED DESCRIPTION:
Pregnancy pathologies can occur from implantation until childbirth. Clinical and scientific investigators are interested in the study of the mechanisms of development of these pathologies and aim to develop therapies to treat them.

The investigators need to collect samples, especially placental samples, following abortions, term, and premature deliveries. Abortions will allow investigators to have non-pathological placental material up to 13 weeks. This material will serve as a reference for understanding the histological changes that occur in normal placentas collected at term of pregnancy. The latter, will in turn, be compared with the placentas collected during premature deliveries. Also, the abortion product will be cultivated in an environment mimicking the pathology of preeclampsia. This study will allow investigators to advance the understanding of the pathophysiological mechanisms of the placenta.

The investigators are internationally recognized for its research on these thematic.

ELIGIBILITY:
Inclusion Criteria:

Adult women

* Admitted to the CHUGA for a birth or an abortion.
* Pregnant women consenting to the collection of their fetal placenta membranes, during premature deliveries or at term of pregnancy OR Women performing an abortion consenting to the collection of their abortion products.
* Having signed a consent
* Affiliated with social security

Exclusion Criteria:

* Placental sample or abortion product unavailable (not collected or necessary for treatment).
* Patient with known positive HIV or Hepatitis B or Hepatitis C serology or at risk according to the infectious safety criteria applied by the EFS.
* hemoglobin <7d / dL or hemoglobin <10g / dL if she suffers from a cardio-respiratory pathology).
* Patient protected by law (minor, hospitalized under duress, subject to a legal protection measure by guardianship or curatorship, deprived of liberty by judicial or administrative decision)

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study will include normal and pathological pregnant women from first to third trimester. A finaliser
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-06 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
To better characterize pregnancy pathologies from implantation to childbirth | Analyses will be performed on each collected sample. The measurement is assessed for up to 6 hours
  Comparison of the frequencies (in percentage) of the histological differences of the placenta and its appendages in patients with pathological and normal pregnancies (histological differences of normal pregnancies versus pathological pregnancies.

SECONDARY OUTCOMES:
Link between the frequencies of histological aberrations and worsening of the pathology | Assessement of the link between the frequencies of histological aberrations and worsening of the pathology will be assessed on the final cohort; This will take up to 3 hours for each aberration.
  Comparison of the severity of the pathology according to the frequencies of aberrations

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Hoffmann, MD PHD, Principal Investigator — Grenoble hospital; Nadia Alfaidy, PhD, Study Director — INSERM U1292

IPD SHARING:
Plan to Share IPD: No